CLINICAL TRIAL: NCT03838965
Title: The Effects of Labor Stages and Interventions on Hemodynamic Measures During and After Childbirth (Epidural, Rupture of Membranes, Cesarean Sections and Preeclampsia) With Noninvasive Sensors.
Brief Title: The Effects of Labor Stages and Interventions on Hemodynamic Measures During & After Childbirth With Noninvasive Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0101-18-HYMC
Record Dates: First submitted 2019-01-30; First posted 2019-02-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Rupture of Membranes; Premature; Cesarean Section; Infection; Preeclampsia
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Infections; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biobeat sensor (Experimental)
  Interventions: Device: biobeat sensor

INTERVENTIONS:
Device: biobeat sensor — biobeat sensor is a noninvasive sensor of the the hymodynamic measures during the childbirth and after 24 hours.

SUMMARY:
The Effects of Labor Stages and Interventions on Hemodynamic Measures During and After Childbirth ( Epidural, Rupture Membranses Cesarean Sections and Preeclampsia) With Noninvasive Sensors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman between 18-45 years old
* with non cardiovascular disease

Exclusion Criteria:

* woman with a cardiovascular disease
* woman who don't agree to participate in the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
biobeat sensor is a noninvasive sensor of the the hymodynamic measures during the childbirth | 24 hours
  biobeat sensor is a noninvasive sensor of the the hymodynamic measures during the childbirth

SECONDARY OUTCOMES:
biobeat sensor is a noninvasive sensor of the the hymodynamic measures after 24 hours of the childbirth | 24 hours
  biobeat sensor is a noninvasive sensor of the the hymodynamic measures after 24 hours of the childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Atsmon, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No